CLINICAL TRIAL: NCT04573244
Title: A Prospective Feasibility Study to Explore the Utility of Using a Smartphone Camera to Monitor Blood Hemoglobin Levels in Children and Adolescents
Brief Title: Hemoglobin Easy Measurement With Optical Artificial Intelligence
Acronym: HEMO-AI
Status: Completed | Type: Observational
Sponsor: MYOR Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EMC 150-20
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-11

CONDITIONS: Hemoglobin; Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood hemoglobin levels are an extremely important measure for a large swath of medical procedures as they reflect the oxygen-carrying capacity of human blood. The gold standard measure for blood hemoglobin levels involve a venous blood draw followed by a laboratory-based complete blood count (CBC), a process which is both painful and time consuming. To date, various methodologies have been tested to either expediate the process or provide a non-invasive alternative. There remains a need to provide a quick, pain-free/non-invasive and accurate modality to measure blood hemoglobin levels. The objective of this study is to determine whether computer vision technologies can be applied to fingernail images captured via a smartphone camera to quantify blood hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

1. A patient aged 6 months to 18 years.
2. A patient who has undergone a venous blood draw for a CBC since being admitted to the PED no more than 6 hours prior to study enrollment.
3. Parents or legal guardian provide informed written consent.

Exclusion Criteria:

1. Patient has subungual hematoma, nail bed lacerations or avulsion injuries on both hands.
2. Patient has total leukonychia.
3. Patient has nail polish applied on fingernails.
4. Patient has nailbed darkening or discoloration due to medication.
5. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient safety.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to the Pediatric Department, Pediatric Emergency Department (PED) or Pediatric Hematology Unit (PHU) who have undergone a CBC
Sampling Method: Non-Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
To determine whether computational learning methods can be applied to fingernail images captured via a smartphone camera to quantify blood hemoglobin levels. | 6 months
  Evaluated using the hemoglobin portion of a conventional complete blood count (CBC)

SECONDARY OUTCOMES:
To determine whether computational learning methods can be applied to fingernail images captured via a smartphone camera to screen for anemia as defined by the WHO | 6 months
  Evaluated using the hemoglobin portion of a conventional complete blood count (CBC). Anemia cutoff for children aged 6 months to 6 years = 11 g/dL and for children aged 6-14 years = 12 g/dL.
To determine whether computational learning methods can be applied to fingernail images captured via a smartphone camera to quantify other elements of the CBC | 6 months
  Evaluated using the hemoglobin portion of a conventional complete blood count (CBC)

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Moshe Chayen, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon D, Hoffman J, Gamrasni K, Barlev Y, Levine A, Landau T, Shpiegel R, Lahad A, Koren A, Levin C, Naor O, Lee H, Liu X, Patel S, Chayen G, Brandwein M. Artificial intelligence-enabled non-invasive ubiquitous anemia screening: The HEMO-AI pilot study on pediatric population. Digit Health. 2024 Dec 5;10:20552076241297057. doi: 10.1177/20552076241297057. eCollection 2024 Jan-Dec. PMID 39640961